CLINICAL TRIAL: NCT00815659
Title: Open-labelled, Single Arm, Phase IV Clinical Study to Evaluate the Impact of Rosuvastatin on Lipid Levels in Patients With Metabolic Syndrome (EFFORT)
Brief Title: Effect of Crestor (Rosuvastatin) on Lipid Levels in Patients With Metabolic Syndrome
Acronym: EFFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00079
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2011-07-04 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Metabolic Syndrome
Keywords: plasma lipid profile; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental): medication start dose is 10mg. After 6 weeks of treatment will be force-titrated to 20mg.
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — medication start dose is 10mg. After 6 weeks of treatment will be force-titrated to 20mg.
  Other Names: CRESTOR

SUMMARY:
The primary objective is to evaluate the efficacy of rosuvastatin therapy on plasma lipid profile (Low Density Lipoprotein (LDL), High-Density Lipoprotein (HDL), total cholesterol, triglyceride) in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome (according to National Cholesterol Education Program (NCEP) Adenosine triphosphate (ATP) Ill criteria)
* LDL-Cholesterol > 130mg/dl
* HDL-Cholesterol < 40mg/dl in males and <50mg/dl in females
* Triglycerides < 400 mg/dl

Exclusion Criteria:

* With a concomitant coronary disease
* Currently under statin therapy or previously treated with statins within the last 6 months

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ural, MD, Prof, Principal Investigator — Kocaeli University Faculty of Medicine Cardiology Dept
Locations (6):
- Turkey (Türkiye) (6):
  - Research site, Ankara, Besevler
  - Research site, Kayseri, Erciyes
  - Research site, Istanbul, Haseki
  - Research site, Kocaeli, Umuttepe
  - Research Site, Izmir
  - Research Site, Trabzon

RESULTS

PARTICIPANT FLOW:
Groups:
- Crestor: Rosuvastatin 10 mg/day for 6 weeks, then 20 mg/day for 6 more weeks
Period: Overall Study
Arm/Group | Crestor
Started | 97
Completed | 74
Not Completed | 23
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Crestor
Number analyzed (Participants) | 97
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Basal HDL-cholesterol Level
Description: HDL-cholesterol levels before (mean of visit 1 - screening and Visit 2 - enrollment)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/dL | 39.5 (6.5)

2. Primary Outcome: HDL-cholesterol Level After 3 Months of Rosuvastatin Treatment
Description: HDL- cholesterol levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) HDL levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/dL | 43.4 (9.8)

3. Primary Outcome: Basal LDL-cholesterol Level
Description: LDL-cholesterol levels before (mean of visit 1 - screening and Visit 2 - enrollment)
Time Frame: Baseline
Population: Baseline LDL levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/dL | 165.5 (32.0)

4. Primary Outcome: LDL-cholesterol Level After 3 Months of Rosuvastatin Treatment
Description: LDL- cholesterol levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) LDL levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/dL | 98.3 (44.8)

5. Primary Outcome: Basal Total Cholesterol Level
Description: Baseline
Time Frame: Total cholesterol levels before (mean of visit 1 - screening and Visit 2 - enrollment)
Population: Baseline total cholesterol levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/dL | 236.5 (38.2)

6. Primary Outcome: Total Cholesterol Level After 3 Months of Rosuvastatin Treatment
Description: Total cholesterol after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) total cholesterol levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/dL | 166.2 (47.7)

7. Primary Outcome: Basal Triglyceride Level
Description: Triglyceride levels before (mean of visit 1 - screening and Visit 2 - enrollment)
Time Frame: Baseline
Population: Baseline triglyceride levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/dL | 195.1 (65.3)

8. Primary Outcome: Triglyceride Level After 3 Months of Rosuvastatin Treatment
Description: Triglycerides after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) triglyceride levels of participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/dL | 153.1 (76.8)

9. Primary Outcome: Number of Patients Who Reached Target Level of LDL-cholesterol After 3 Months of Rosuvastatin Treatment
Description: Number of patients who reached target level of LDL-cholesterol after 3 months of rosuvastatin treatment. Target level: LDL-cholesterol: <100 mg/dL; HDL-cholesterol: For males >40 mg/dL, for females >50 mg/dL; non-HDL-cholesterol: <130 mg/dL
Time Frame: 3 months (from enrollment to last visit)
Population: LDL cholesterol levels < 100 mg/dL, calculated over patients with lipid measurement performed at both visits
Measure: Number; unit: Participants
Arm/Group | Crestor
Number analyzed (Participants) | 65
Participants | 48

10. Primary Outcome: Number of Patients Who Reached Target Level of HDL-cholesterol After 3 Months of Rosuvastatin Treatment
Description: Number of patients who reached target level of HDL-cholesterol after 3 months of rosuvastatin treatment
Time Frame: 3 months (from enrollment to last visit)
Population: HDL cholesterol target levels for males >40 mg/dL, for females > 50 mg/dL, calculated over patients with lipid measurement performed at both visits
Measure: Number; unit: Participants
Arm/Group | Crestor
Number analyzed (Participants) | 66
Participants | 39

11. Primary Outcome: Number of Patients Who Reached Target Level of Non-HDL-cholesterol After 3 Months of Rosuvastatin Treatment
Description: Number of patients who reached target level of non-HDL-cholesterol after 3 months of rosuvastatin treatment
Time Frame: 3 months (from enrollment to last visit)
Population: Non-HDL cholesterol target levels <130 mg/dL, calculated over patients with lipid measurement performed at both visits
Measure: Number; unit: Participants
Arm/Group | Crestor
Number analyzed (Participants) | 66
Participants | 51

12. Secondary Outcome: Basal Interleukin 1 (IL-1) Level
Description: IL-1 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline IL-1 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
pg/mL | 4.1 (2.3)

13. Secondary Outcome: Interleukin 1 (IL-1) Level After 3 Months of Rosuvastatin Treatment
Description: IL-1 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) IL-1 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
pg/mL | 4.1 (2.2)

14. Secondary Outcome: Basal Interleukin 6 (IL-6) Level
Description: IL-6 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline IL-6 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
pg/mL | 2.6 (2.1)

15. Secondary Outcome: Interleukin 6 (IL-6) Level After 3 Months of Rosuvastatin Treatment
Description: IL-6 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) IL-6 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
pg/mL | 2.8 (2.8)

16. Secondary Outcome: Basal Interleukin 8 (IL-8) Level
Description: IL-8 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline IL-8 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
pg/mL | 10.7 (5.1)

17. Secondary Outcome: Interleukin 8 (IL-8) Level After 3 Months of Rosuvastatin Treatment
Description: IL-8 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) IL-8 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
pg/mL | 12.7 (13.3)

18. Secondary Outcome: Basal Interleukin 10 (IL-10) Level
Description: IL-10 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline IL-10 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
pg/mL | 4.2 (2.1)

19. Secondary Outcome: Interleukin 10 (IL-10) Level After 3 Months of Rosuvastatin Treatment
Description: IL-10 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) IL-10 levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
pg/mL | 4.8 (3.9)

20. Secondary Outcome: Basal Tumor Necrosis Factor (TNF) Level
Description: TNF levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline Basal Tumor Necrosis Factor (TNF) levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
pg/mL | 10.8 (5.3)

21. Secondary Outcome: Tumor Necrosis Factor (TNF) Level After 3 Months of Rosuvastatin Treatment
Description: TNF levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) Tumor Necrosis Factor (TNF) levels of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
pg/mL | 12.9 (9.2)

22. Secondary Outcome: Basal High Sensitivity C-reactive Protein (Hs-CRP) Level
Description: hs-CRP levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline High Sensitivity C-reactive protein (Hs-CRP) levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 8.2 (7.3)

23. Secondary Outcome: High Sensitivity C-reactive Protein (Hs-CRP) Level After 3 Months of Rosuvastatin Treatment
Description: hs-CRP levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) High Sensitivity C-reactive protein (Hs-CRP) levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 6.7 (5.6)

24. Secondary Outcome: Basal LDL-3 Level
Description: LDL subfractions are light (LDL1 and 2), intermediate (LDL3) and small dense LDL (LDL 4, 5, 6 and 7). Small dense LDL (sdLDL)-cholesterol that expresses greater atherogenicity than large buoyant LDL. Large LDL particles are the least likely to cause plaque formation, because LDL particles have to be approximately 25 nm in diameter or smaller to penetrate the artery walls. High sdLDL and decreased large HDL fraction are more common in patients with coronary heart disease than in controls
Time Frame: Baseline
Population: Baseline LDL-3 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 15.5 (9.5)

25. Secondary Outcome: LDL-3 Level After 3 Months of Rosuvastatin Treatment
Description: LDL-3 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) LDL-3 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 8.8 (7.9)

26. Secondary Outcome: Basal LDL-4 Level
Description: LDL-4 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline LDL-4 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 7.9 (9.6)

27. Secondary Outcome: LDL-4 Level After 3 Months of Rosuvastatin Treatment
Description: LDL-4 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF(Last Observation Carried Forward) LDL-4 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 3.5 (4.8)

28. Secondary Outcome: Basal LDL-5 Level
Description: LDL-5 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline LDL-5 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 2.7 (7.1)

29. Secondary Outcome: LDL-5 Level After 3 Months of Rosuvastatin Treatment
Description: LDL-5 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) LDL-5 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 1.3 (3.5)

30. Secondary Outcome: Basal LDL-6 Level
Description: LDL-6 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline LDL-6 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 0.5 (2.6)

31. Secondary Outcome: LDL-6 Level After 3 Months of Rosuvastatin Treatment
Description: LDL-6 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) LDL-6 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 0.3 (1.5)

32. Secondary Outcome: Basal LDL-7 Level
Description: LDL-7 levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline LDL-7 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 0.5 (3.0)

33. Secondary Outcome: LDL-7 Level After 3 Months of Rosuvastatin Treatment
Description: LDL-7 levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) LDL-7 levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 0.8 (5.3)

34. Secondary Outcome: Basal Large HDL Subfraction Level
Description: Large HDL subfraction levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline Large HDL subfraction of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 15.0 (6.4)

35. Secondary Outcome: Large HDL Subfraction Level After 3 Months of Rosuvastatin Treatment
Description: Large HDL subfraction levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) Large HDL subfraction levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 17.6 (7.6)

36. Secondary Outcome: Basal Intermediate HDL Subfraction Level
Description: Intermediate HDL subfraction levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline Intermediate HDL subfraction of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 18.9 (5.7)

37. Secondary Outcome: Intermediate HDL Subfraction Level After 3 Months of Rosuvastatin Treatment
Description: Intermediate HDL subfraction levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) Intermediate HDL subfraction levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 19.9 (6.1)

38. Secondary Outcome: Basal Small HDL Subfraction Level
Description: Small HDL subfraction levels before (Visit 2-enrollment)
Time Frame: Baseline
Population: Baseline Small HDL subfraction of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 97
mg/mL | 6.2 (4.2)

39. Secondary Outcome: Small HDL Subfraction Level After 3 Months of Rosuvastatin Treatment
Description: Small HDL subfraction levels after 3 months of rosuvastatin treatment (last observation carried forward; LOCF)
Time Frame: 3 months (from enrollment to last visit)
Population: LOCF (Last Observation Carried Forward) Small HDL subfraction levels of participants
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Crestor
Number analyzed (Participants) | 96
mg/mL | 6.6 (4.6)

40. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of patients with any adverse events in 3 months of rosuvastatin treatment
Time Frame: 3 months (from enrollment to last visit)
Population: Number of patients with any adverse events in 3 months
Measure: Number; unit: Participants
Arm/Group | Crestor
Number analyzed (Participants) | 97
Participants | 24

ADVERSE EVENTS:
Arm/Group | Crestor
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 29/97
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crestor (N=97)
Myalgia (Musculoskeletal and connective tissue disorders) | 2
CK Increased (Investigations) | 2
Dysuria (Infections and infestations) | 2
Pruritus-Allergy-Rash (Skin and subcutaneous tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 1
Allergy (Gastrointestinal disorders) | 1
Dermatoid (Skin and subcutaneous tissue disorders) | 1
Eye Twitching (Eye disorders) | 1
Blood Pressure Increased (Eye disorders) | 1
Weight Increased (Eye disorders) | 1
Leg Cramp (Musculoskeletal and connective tissue disorders) | 1
Leg Swelling (Musculoskeletal and connective tissue disorders) | 1
Cough-Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Liver Function Tests Abnormal (Infections and infestations) | 2
Headache (Skin and subcutaneous tissue disorders) | 4
Acute Pneumonia (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other